CLINICAL TRIAL: NCT00245739
Title: Early Access of TMC114 in Combination With Low-dose Ritonavir (TMC/r)) and Other Antiretrovirals (ARVs) in Highly Treatment Experienced HIV-1 Infected Patients With Limited to no Treatment Options.
Brief Title: TMC114-C226: An Early Access Program to Evaluate the Long-term Safety and Tolerability of TMC114 Combined With a Low Dose of Ritonavir (TMC114/r) With Other Antiretrovirals, for HIV-1 Infected Patients Who Have Failed Multiple Antiretroviral Regimens.
Status: Approved for marketing | Type: Expanded Access
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Other Study IDs: CR006304; TMC114-C226 (Other: Tibotec Pharmaceuticals, Ireland); NCT00613483 (obsolete NCT alias)
Record Dates: First submitted 2005-10-27; First posted 2005-10-28 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-04

CONDITIONS: HIV Infections
Keywords: HIV infections; HIV-1; TMC114; Early access; Highly antiretroviral treatment experienced patients; Anti-retroviral agents
MeSH Terms: conditions — HIV Infections | interventions — Darunavir

INTERVENTIONS:
Drug: TMC-114 — 600/100 mg tablets of TMC114/rtv BID until commercial available to the subject

SUMMARY:
The purpose of this study is to provide early access to TMC114 (a protease inhibitor) for HIV-1 infected patients with limited or no treatment options, who have failed multiple antiretroviral (ARV) regimens, and to evaluate the longer-term safety and tolerability of TMC114/r in combination with other antiretrovirals

DETAILED DESCRIPTION:
This is a program to provide early access to TMC114 (a protease inhibitor) for HIV-1 infected patients, who have failed multiple antiretroviral (ARV) regimens and who are ineligible for participation in any other Tibotec-sponsored HIV trial. Patients need to be at least 3 class experienced (PIs, NRTIs, NtRTIs, NNRTIs or FI), to have previously received 2 different protease inhibitor-based regimens and to not be virologically suppressed on their current regimen. Patients eligible for any other Tibotec sponsored HIV trial but located more than 100 kilometers away from a study site, will be considered eligible for this early access program.

This program will be conducted as an open-label, non-randomized treatment study. Once treatment with TMC114/r in combination with other antiretrovirals (ARVs) has been initiated (baseline visit), patients will follow the recommended visit schedule based on routine clinical care. No other protease inhibitor combinations other than TMC114/r are to be used in this study, except atazanavir (ATV) and indinavir (IDV) may be allowed. Trial medication will be dispensed every 8 weeks. Treatment with TMC114/r will be continued until treatment-limiting toxicity, loss to follow-up, patient's withdrawal, pregnancy, discontinuation of TMC114 development or when TMC114 has become commercially available.

Selected safety and tolerability data, including adverse events will be collected throughout the study. A urine pregnancy test will be repeated at baseline for female patients if more than 4 weeks have passed since the test at screening, and urine pregnancy tests will be performed at all other visits. In addition, data on CD4 count and viral load will be collected over the treatment period according to local standard of care practice, in order to ensure that patients continue to benefit from treatment with TMC114/r. A final/withdrawal visit as well as a post-trial treatment follow-up contact (4 weeks after the final/withdrawal visit) will be performed. Patients will take oral doses of 600 mg of TMC114 twice daily in combination with 100 mg of ritonavir twice daily, in combination with other antiretrovirals.

ELIGIBILITY:
Inclusion Criteria:

* Patient with documented HIV-1 infection
* has limited or no treatment options due to virological failure or intolerance to multiple antiretroviral regimens
* is at least 3 class experienced and has previously received 2 different protease inhibitor-based regimens
* has a CD4 cell count <= 200 cells/mm3
* is not achieving adequate virologic suppression on his/her current regimen and is at risk of clinical or immunologic progression.

Exclusion Criteria:

* Patient has primary HIV-1 infection (unless documented resistance to all currently approved protease inhibitors participated or is currently participating in a trial with TMC114
* Patient used investigational medication within the last 30 days (except for abacavir/lamivudine and tenofovir/emtricitabine fixed dose combinations, and tipranavir)
* Patient suffers from any active clinically significant disease (e.g., cardiac dysfunction, pancreatitis, acute viral infection) or has evidence of active liver disease, liver impairment/dysfunction or cirrhosis irrespective of liver enzyme levels, or has grade 3 or 4 laboratory abnormalities as defined by National Institute of Allergy and Infectious Diseases Division of AIDS (DAIDS) grading scheme
* Female patients that are pregnant or breast-feeding, or of childbearing potential without using effective non-hormonal birth control methods or not willing to continue practicing these birth control methods from screening until the last trial related activity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited
Locations (394):
- United States (202):
  - Anniston, Alabama
  - Birmingham, Alabama
  - Mesa, Arizona
  - Phoenix, Arizona
  - Tucson, Arizona
  - Anaheim, California
  - Bakersfield, California
  - Baldwin Park, California
  - Beverly Hills, California
  - Carmichael, California
  - Fontana, California
  - Fountain Valley, California
  - French Camp, California
  - Glendale, California
  - Harbor City, California
  - Hayward, California
  - Loma Linda, California
  - Long Beach, California
  - Los Angeles, California
  - Los Angles, California
  - Newport Beach, California
  - Oakland, California
  - Palm Springs, California
  - Palo Alto, California
  - Panorama City, California
  - Paramount, California
  - Richmond, California
  - Salinas, California
  - San Diego, California
  - San Diego, La Jolla, California
  - San Francisco, California
  - San Mateo, California
  - San Rafael, California
  - Santa Ana, California
  - Santa Clara, California
  - Santa Clarita, California
  - Santa Rosa, California
  - Stanford, California
  - Sunnyvale, California
  - Tarzana, California
  - Ukiah, California
  - West Hollywood, California
  - Woodland Hills, California
  - Denver, Colorado
  - Glastonbury, Connecticut
  - Hartford, Connecticut
  - New Haven, Connecticut
  - Norwalk, Connecticut
  - Norwich, Connecticut
  - Stanford, Connecticut
  - Vernon Rockville, Connecticut
  - Washington D.C., District of Columbia
  - Boynton Beach, Florida
  - Brandon, Florida
  - Fort Lauderdale, Florida
  - Fort Laudersale, Florida
  - Fort Myers, Florida
  - Hollywood, Florida
  - Jacksonville, Florida
  - LaBelle, Florida
  - Melbourne, Florida
  - Miami, Florida
  - Miami Beach, Florida
  - North Miami Beach, Florida
  - North Palm Beach, Florida
  - Orlando, Florida
  - Plantation, Florida
  - Port Saint Lucie, Florida
  - Safety Harbor, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - Vero Beach, Florida
  - West Palm Beach, Florida
  - Winter Park, Florida
  - Atlanta, Georgia
  - Augusta, Georgia
  - Austell, Georgia
  - Decatur, Georgia
  - Jesup, Georgia
  - Macon, Georgia
  - Marietta, Georgia
  - Riverdale, Georgia
  - Tucker, Georgia
  - Honolulu, Hawaii
  - Kahului, Hawaii
  - Kapaa, Hawaii
  - Boise, Idaho
  - Chicago, Illinois
  - Decatur, Illinois
  - Granite City, Illinois
  - Joliet, Illinois
  - Rockford, Illinois
  - Round Lake Beach, Illinois
  - Springfield, Illinois
  - Topeka, Kansas
  - Henderson, Kentucky
  - Paducah, Kentucky
  - New Orleans, Louisiana
  - Bangor, Maine
  - Lewiston, Maine
  - Monmouth, Maine
  - Portland, Maine
  - Baltimore, Maryland
  - Bethesda, Maryland
  - Elkton, Maryland
  - Silver Spring, Maryland
  - Boston, Massachusetts
  - Cambridge, Massachusetts
  - Springfield, Massachusetts
  - Berkley, Michigan
  - Detroit, Michigan
  - Grosse Pointe Woods, Michigan
  - Marquette, Michigan
  - Minneapolis, Minnesota
  - Greenwood, Mississippi
  - Columbia, Missouri
  - Kansas City, Missouri
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Lebanon, New Hampshire
  - East Orange, New Jersey
  - Galloway, New Jersey
  - Hackensack, New Jersey
  - Hamilton, New Jersey
  - Hoboken, New Jersey
  - Jersey City, New Jersey
  - Long Branch, New Jersey
  - Maplewood, New Jersey
  - Neptune City, New Jersey
  - Newark, New Jersey
  - Perth Amboy, New Jersey
  - Somers Point, New Jersey
  - Voorhees Township, New Jersey
  - West Orange, New Jersey
  - Westfield, New Jersey
  - Albuquerque, New Mexico
  - Albany, New York
  - Briarcliff, New York
  - Bronxville, New York
  - Brooklyn, New York
  - Flushing, New York
  - Harris, New York
  - Manhasset, New York
  - Mount Vernon, New York
  - New York, New York
  - Rochester, New York
  - Syracuse, New York
  - The Bronx, New York
  - Valhalla, New York
  - Yonkers, New York
  - Asheville, North Carolina
  - Chapel Hill, North Carolina
  - Greensboro, North Carolina
  - Greenville, North Carolina
  - Huntersville, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Akron, Ohio
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Dayton, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Allentown, Pennsylvania
  - Easton, Pennsylvania
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - West Reading, Pennsylvania
  - Providence, Rhode Island
  - Charleston, South Carolina
  - Columbia, South Carolina
  - West Columbia, South Carolina
  - Hermitage, Tennessee
  - Johnson City, Tennessee
  - Knoxville, Tennessee
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Bryan, Texas
  - Dallas, Texas
  - El Paso, Texas
  - Fort Worth, Texas
  - Galveston, Texas
  - Harlingen, Texas
  - Houston, Texas
  - Lackland City, Texas
  - Longview, Texas
  - San Antonio, Texas
  - Annandale, Virginia
  - Charlottesville, Virginia
  - Fairfax, Virginia
  - Hampton, Virginia
  - Newport News, Virginia
  - Norfolk, Virginia
  - Portsmouth, Virginia
  - Richmond, Virginia
  - Seattle, Washington
  - Eau Claire, Wisconsin
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Belgium (8):
  - Antwerp
  - Bruges
  - Brussels
  - Charleroi
  - Ghent
  - Leuven
  - Liège
  - Yvoir
- Canada (18):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Moncton, New Brunswick
  - Halifax, Nova Scotia
  - Hamilton, Ontario
  - Kingston, Ontario
  - London, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Whitby, Ontario
  - Windsor, Ontario
  - Montreal, Quebec
  - Rouyn-Noranda, Quebec
  - Ste-Foy, Quebec
  - Vancouver
  - Vancouver British
- Prague, Czechia
- Denmark (5):
  - Aalborg
  - Aarhus
  - Copenhagen
  - Hvidovre
  - Odense
- Germany (35):
  - Aachen
  - Berlin
  - Bochum
  - Bonn
  - Bremen
  - Chemnitz
  - Cologne
  - Dortmund
  - Dresden
  - Düsseldorf
  - Erlangen
  - Essen
  - Frankfurt
  - Freiburg im Breisgau
  - Giessen
  - Hamburg
  - Hanover
  - Kiel
  - Koblenz
  - Konstanz
  - Kÿln
  - Leipzig
  - Mainz
  - Mannheim
  - Munich
  - München
  - Münster
  - Nuremberg
  - Osnabrück
  - Regensburg
  - Saarbrücken
  - Salzgitter
  - Stuttgart
  - Wuppertal
  - Würzburg
- Greece (3):
  - Athens
  - Piraeus
  - Thessalonikis
- Budapest, Hungary
- Luxembourg, Luxembourg
- Malaysia (3):
  - Ipoh
  - Kuala Lumpur
  - Pulau Pinang
- Mexico (9):
  - Col Tacuba
  - Guadalajara
  - Mex Ctity
  - Mexico City
  - México
  - Monterrey Nuevo León
  - Oaxaca City
  - Puebla City
  - Veracruz
- Netherlands (12):
  - Alkmaar
  - Amsterdam
  - Arnhem
  - Eindhoven
  - Enschede
  - Groningen
  - Leiden
  - Maastricht
  - Nijmegen
  - Rotterdam
  - The Hague
  - Tilburg
- Puerto Rico (3):
  - Ponce Pr
  - Rio Piedras Pr
  - San Juan
- Russia (12):
  - Kazan'
  - Krasnodar
  - Moscow
  - Nizhny Novgorod
  - Novosibirsk Region
  - Rostov-on-Don
  - Saint Petersburg
  - Smolensk
  - Tver'
  - Volgograd
  - Voronezh
  - Yekaterinburg
- Ljubljana, Slovenia
- Spain (56):
  - A Coruña
  - Alicante
  - Badajoz
  - Barakaldo Vizcaya S/N
  - Barcelona
  - Bilbao
  - Calella (Barcelona)
  - Castellon
  - Cáceres
  - Córdoba
  - Cuenca
  - Donostia Guipuzcoa
  - El Palmar Murcia N/A
  - Elche
  - Figueres
  - Fuenlabrada
  - Gijon Asturias
  - Girona
  - Granada
  - Guadalajara
  - Huelva
  - Huesca
  - Ibiza Town
  - Jérez
  - Las Palmas de Gran Canaria
  - León
  - Lleida
  - Logroño
  - Madrid
  - Manresa
  - Maó
  - Málaga
  - Murcia
  - Oviedo
  - Palma de Mallorca
  - Palma de Mallorca Illes Balear
  - Pamplona
  - Puerto Real
  - Sabadell
  - Salamanca
  - San Cristóbal de La Laguna
  - Santa Cruz de Tenerife
  - Santander
  - Santiago de Compostela
  - Seville
  - Tarragona
  - Terrassa
  - Valencia
  - Valladolid
  - Vic
  - Vigo
  - Villafranca Del Penedes
  - Vitoria-Gasteiz
  - Vizcaya N/A
  - Zamora
  - Zaragoza
- Sweden (5):
  - Gothenburg
  - Linköping
  - Malmo
  - Stockholm
  - Uppsala
- Switzerland (11):
  - Aarau
  - Basel
  - Bern
  - Bruderholz
  - Chur
  - Geneva
  - Lausanne
  - Lugano
  - Sankt Gallen
  - Zurich
  - Zurich Zh
- Taiwan (4):
  - Kaohsiung City
  - Kaohsiung County
  - Taipei
  - Taoyuan District
- Bangkok, Thailand
- Turkey (Türkiye) (2):
  - Ankara
  - Istanbul
- Caracas, Venezuela